CLINICAL TRIAL: NCT05016492
Title: Interactive Digital Game for Improving Visual Perceptual Defects in Children With Developmental Disability: Evaluation of Efficacy and User Satisfaction
Brief Title: Interactive Digital Game for Improving Visual Perceptual Defects in Children With Developmental Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMUHIRB-SV(II)-20150090
Record Dates: First submitted 2021-08-17; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Developmental Disability
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Digital game group (Experimental): The digital game group received the standard 4-week course of rehabilitation but with an additional 30-min interactive digital game training session per week.
  Interventions: Device: Visual-perceptual interactive game system; Behavioral: standard rehabilitation
- Standard rehab group (Active Comparator): The standard rehab group received the standard 4-week course of rehabilitation delivered in one 30-min session per week.
  Interventions: Behavioral: standard rehabilitation

INTERVENTIONS:
Device: Visual-perceptual interactive game system — Subjects received 30-min interactive digital game training session per week. The game system contain 7 skills training, each of which was named according to the corresponding TVPS-3.
  Arms: Digital game group
Behavioral: standard rehabilitation — Subjects received the standard 4-week course of rehabilitation delivered in one 30-min session per week. The course of rehabilitation included: sensory integration therapy, cognitive function training and visual perception/auditory attention training.

SUMMARY:
Visual perceptual defects in children can negatively affect their activities of daily living.The aims of this study were to develop and evaluate an interactive digital game system for correcting visual perceptual defects and to evaluate the effectiveness of the proposed system.

ELIGIBILITY:
Inclusion Criteria:

* Record of developmental disability diagnosis
* Ability to understand instructions
* TVPS-3 score lower than 25% of the norm reference and diagnosis of visual perceptual defect
* Test of Nonverbal Intelligence-3rd Edition score higher than 70

Exclusion Criteria:

* Did not follow or understand the instructions for participating in the study
* Had severe defects in vision, hearing, etc.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2016-05-24 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2017-05-23 (Actual)

PRIMARY OUTCOMES:
Test of Visual Perceptual Scale-3(TVPS-3) | 4 weeks
  TVPS-3 is a standardized and norm-referenced task for children age 4-13 years that uses a response format suitable for all children, including those with disabilities. It includes subtasks of visual discrimination, visual memory, visual-spatial relationships, form constancy, visual sequential memory, figure ground, and visual closure (Martin et al., 2006). Each of the seven subtests has 16 items of varying difficulty. Therefore, the test has 112 total questions.
User satisfaction survey | 4 weeks
  The 20-item questionnaire content was divided into five themes: perceived ease of use (6 questions), perceived usefulness (4 questions), perceived joyfulness (4 questions), satisfaction (3 questions), and continued use (3 questions). Questionnaire items were answered on a Likert scale from 1 (completely disagree) to 5 (completely agree).
Test of the visual-perceptual interactive game system | 4 weeks
  The digital game test had 7 subtests, and each subtest had 10 questions. Based on the seven-item rules of TVPS-3, 1 point was assigned to each question, for a score of 10 points for each subtest, and a total score of 70.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Wu WL, Huang YL, Liang JM, Chen CH, Wang CC, Ho WH. Interactive Digital Game for Improving Visual-Perceptual Defects in Children With a Developmental Disability: Randomized Controlled Trial. JMIR Serious Games. 2022 Apr 15;10(2):e34756. doi: 10.2196/34756. PMID 35436215